CLINICAL TRIAL: NCT05946629
Title: A Prospective Randomized Single-Blind Multicenter Study to Assess the Safety and Effectiveness of the SELUTION SLR™ 014 PTCA Drug Eluting Balloon in the Treatment of Subjects With De Novo Coronary Lesions in Small Vessels
Brief Title: SELUTION 4 De Novo Small Vessel IDE Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.A. Med Alliance S.A. (Industry)
Collaborators: NAMSA (Other); Cordis US Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SEL-003-2021
Record Dates: First submitted 2023-06-30; First posted 2023-07-14 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease
Keywords: CAD; DCB; DEB; NSTEMI; Stable Angina; Chronic Coronary Syndrome; CCS; Drug Coated Balloons; Drug Eluting Balloons; Small Vessels; SELUTIONSLR; Sirolimus
MeSH Terms: conditions — Coronary Artery Disease; Non-ST Elevated Myocardial Infarction; Angina, Stable | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Single-Blind Randomized Control Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The randomized trial is a single-blind study. The physician performing the index procedure as well as study site personnel present at the index procedure will not be blinded, however every effort will be made to maintain blinding for the following:
  * Subjects and their families
  * Site personnel involved in conducting study assessments during follow-up Unblinding will only occur to protect subject rights, welfare, or well-being. The angiographic and pK substudy cohorts will not be blinded.
  The Clinical Events Committee (CEC) will be blinded to the treatment arm during the adjudication process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- SELUTION SLR 014 PTCA DEB (Experimental): SELUTION Sustained Limus Release (SLR) 014 Percutaneous Transluminal Coronary Angioplasty (PTCA) Drug Eluting Balloon (DEB)
  The SELUTION SLR 014 PTCA DEB is a minimally invasive, single use and sterile Sirolimus coated PTCA balloon catheter.
  The SELUTION SLR 014 PTCA DEB is available with balloon diameters from 2.0 to 3.0 mm and lengths of 15 to 40 mm for the purpose of the De Novo IDE trial
  Interventions: Device: PCI with SELUTION SLR DCB
- Control Treatment (Active Comparator): any FDA approved "limus-based" Drug Eluting Stent, as per standard institutional practice
  Interventions: Device: PCI with FDA approved "-limus" DES

INTERVENTIONS:
Device: PCI with SELUTION SLR DCB — After target lesion pre-dilatation and preparation , a SELUTION SLR 014 PTCA DEB study device should be selected with nominal diameter equal to the RVD of the target lesion (1:1 ratio) and length that allows approximately 2.00 mm longer than the proximal and distal edges of the target lesion (defined as the proximal and distal extent of predilation). If IVUS is performed to assess RVD, and DEB upsizing is deemed clinically necessary for optimal results, a maximum nominal DEB diameter of 3.0 mm is permitted. The SELUTION SLR 014 PTCA DEB should then be delivered, positioned in and deployed per instructions per use. The balloon should be inflated for 60 seconds provided that the patient can tolerate this duration. The minimum inflation time is 30 seconds.
  Arms: SELUTION SLR 014 PTCA DEB
Device: PCI with FDA approved "-limus" DES — For subjects randomized to the control group (DES), the treating physician will choose an FDA cleared DES and follow lesion preparation and stent deployment according to the Instructions per use (IFU) and institutional practices.
  The DES should be sized per IFU with respect to the vessel RVD. The use of IVUS or OCT is encouraged to guide optimal stent placement and assess final results. After DES deployment, additional balloon inflations should be performed as needed to obtain < 30% residual diameter stenosis and resolve proximal or distal edge dissections greater than or equal to NHLBI grade B.
  Arms: Control Treatment

SUMMARY:
Prospective, randomized controlled, single-blind, multicenter, clinical trial to demonstrate the safety and efficacy of the SELUTION SLR 014 PTCA DEB for treatment of de novo lesions in small coronary vessels, defined as reference vessel diameter (RVD) of 2.00 mm to 2.75 mm, in support of a pre-market approval (PMA) application to the United States (US) FDA.

The Study will enroll up to 910 randomized subjects, up to 30 subjects in a parallel angiographic substudy, and up to 20 subjects in a parallel pharmacokinetic (pK) substudy, at up to 80 sites in the US, Canada, Brazil, Japan and Europe. A minimum of 50% of the subjects will be enrolled in the US.

DETAILED DESCRIPTION:
Prospective, randomized controlled, single-blind, multicenter, clinical trial

The study will enroll up to 910 randomized subjects, up to 30 subjects in a parallel angiographic substudy, and up to 20 subjects in a parallel pharmacokinetic (pK) substudy, at up to 80 sites in the US, Canada, Brazil, Japan and Europe. A minimum of 50% of the subjects will be enrolled in the US.

Subjects who present with chronic coronary syndrome (CCS), unstable angina or stabilized non-ST elevation myocardial infarction (NSTEMI) with an indication for percutaneous coronary intervention (PCI) with planned intervention for de novo lesions in small coronary vessels (RVD 2.00 mm to 2.75 mm) and meeting all eligibility criteria will be randomized 1:1 to treatment of the identified target lesion with either the SELUTION SLR 014 PTCA DEB or contemporary DES.

Randomized Cohort:

* Intervention (DEB Strategy): Subjects randomized to the SELUTION SLR 014 PTCA DEB arm will receive lesion preparation according to the 3rd drug coated balloon (DCB) consensus (optimal balloon angioplasty with adjunct treatment using high-pressure balloon, intravascular lithotripsy, laser, rotational or orbital atherectomy, cutting or scoring balloon at the discretion of the operator as needed to reduce diameter stenosis to ≤ 30%). Subjects with lesions that are then best treated by provisional stenting (flow-limiting dissection, residual stenosis > 30%) will receive a DES instead of the SELUTION DEB but remain in the SELUTION DEB group (intention to treat analysis). The DEB should not be used after DES implant.
* Control (DES): Subjects randomized to the DES arm will receive treatment using any FDA approved "limus-based" DES, as per standard institutional practice.

Angiographic Substudy:

The angiographic substudy is a parallel registry consisting of up to 30 additional consecutive subjects meeting all eligibility criteria treated with the SELUTION DEB recruited at select study sites. These subjects will undergo angiography at 12 months post-procedure. Clinical follow-up will not extend beyond 12 months in this cohort.

Pharmacokinetic (pK) Substudy:

The pKsubstudy is a parallel registry consisting of up to 20 additional consecutive subjects meeting all eligibility criteria treated with the SELUTION DEB recruited at select study sites. This study will be conducted under an approved substudy protocol and will include blood draws at regular intervals to characterize the pK plasma profile of sirolimus.

Primary Endpoint:

Target lesion failure (TLF), defined as the composite of cardiac death, target-vessel myocardial infarction (MI) or clinically-driven target lesion revascularization (TLR) at 12 months. MI includes spontaneous (Type 1) MI using the 4th Universal Definition of Myocardial Infarction (UDMI) and peri-procedural MI using the Society for Cardiac Angiography and Intervention (SCAI) definition.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Inclusion Criteria

Subjects must meet all of the following clinical criteria to participate in the trial:

1. Subject is ≥ 18 years (or the minimum legal age as required by local regulations).
2. Female subjects of childbearing potential must have a negative pregnancy test ≤ 7 days before the procedure or are using a contraceptive device or drug.
3. Subject presents with chronic coronary syndromes [CCS] (manifest as documented angina or positive functional testing), unstable angina or stabilized non-ST elevation myocardial infarction (NSTEMI) (biomarkers stabilized or down trending) with an indication for PCI and planned intervention.
4. Subject can tolerate dual antiplatelet therapy with aspirin, plus either Clopidogrel, Prasugrel, or Ticagrelor. (Note: For subjects requiring oral anticoagulation, aspirin may be omitted based on investigator discretion).
5. Subject has life expectancy > 1 year in the opinion of the investigator.
6. Subject is willing and able to provide informed consent and comply with study procedures and required follow-up evaluations.

PK Sub- Study Inclusion Criteria:

Subjects must meet all of the main protocol inclusion criteria to participate in the PK sub-study. Subjects must also meet the following additional PK sub-study inclusion criteria:

1. Subject is willing and able to provide informed consent for the PK sub-study and comply with the PK sub-study procedures and required follow-up evaluations.

Imaging Inclusion Criteria

Subject's target lesion(s) must meet all of the following angiographic criteria for the subject to participate in the trial:

1. A single, target lesions that meet criteria can be treated in a single vessel. No non-target lesions can be treated within the target vessel in the index procedure. Non-target lesions within the target vessel can be staged for treatment > 30 days from the index procedure.
2. Up to two (2) non-target lesions in up to two (2) non-target vessels may be treated, but successful PCI of the non-target lesions must be completed before randomization and treatment of the target lesion.
3. Target lesion is ≤ 36 mm in length.
4. Target lesion has diameter stenosis > 50% and ≤ 99% with distal flow at least thrombolysis in myocardial infarction (TIMI) 2.
5. Target vessel has RVD of ≥ 2.00 mm and ≤ 2.75 mm [by visual assessment].
6. Target lesion is within a native coronary artery or major branch.
7. A target lesion within a bifurcation is allowed only if a single vessel (either main vessel or side branch) is to be treated.
8. The identified target lesion has high probability for successful treatment with approved pre-treatment techniques and DEB alone based on Investigator assessment.

Exclusion Criteria:

* Clinical Exclusion Criteria

Subjects who meet any of the following clinical criteria will be excluded from the trial:

1. Subject with known hypersensitivity or allergy to Sirolimus or its analogues.
2. Subject presents with NSTEMI and rising biomarkers, or ongoing chest pain or is hemodynamically instable.
3. Subject with history of ST-elevation myocardial infarction (STEMI) within 30 days of the index procedure.
4. Subject with planned major surgery within 30 days following the index procedure.
5. Subject with planned treatment of lesion involving aorto-ostial location.
6. Subject with PCI of a non-target vessel within ± 30 days of the index procedure.
7. Subject with history (within 6 months prior to index procedure) of New York Heart Association (NYHA) class III or IV heart failure.
8. Subject with history of active peptic ulcer or gastrointestinal bleeding within 6 months of the index procedure or other inability to comply with the recommended duration of dual antiplatelet therapy (DAPT).
9. Subject is pregnant, breast-feeding or a woman of childbearing potential who plans pregnancy up to 1 year following index procedure.
10. Subjects with current documented left ventricular ejection fraction (LVEF) < 30%.
11. Subject is considered not able to tolerate at least 30 seconds of coronary occlusion for the target lesion treated.
12. Subjects is currently participating in another investigational drug or device study that has not completed primary endpoint follow-up.
13. Subject with definite clinically active COVID-19 infection defined as a positive COVID test within 24 hours of index procedure.
14. Subject has chronic renal insufficiency (dialysis dependent, or glomerular filtration rate [GFR] ≤ 30 ml/min/1.73 m2 within 30 days of index procedure) or had undergone renal transplantation.

PK Sub-Study Exclusion Criteria:

Subjects must meet none of the main protocol exclusion criteria to participate in the PK sub-study. Subjects will be excluded if any of the following additional PK sub-study exclusion criteria are met:

1. Any limus family (Zotarolimus, Everolimus, Sirolimus etc.) eluting device has been placed/used in any part of the body within 3 months prior to the index procedure including non-target lesion(s) treated during the index procedure.
2. Planned intervention with any limus family (Zotarolimus, Everolimus, Sirolimus etc.) eluting device anywhere in the body within 6 months after the index procedure. Note: staged procedures >30 days after index procedure (Exclusion #6 of the main protocol) are permitted only in the main protocol, and are not permitted in this PK sub-study.
3. The subject is taking or has taken within the last 3 months any limus family medication(s) for any reason.
4. Subject is concurrently enrolled in the main protocol angiographic registry.
5. Subjects who are taking strong CYP3A4 Inhibitors within 14 days before the index procedure or plan to take the strong inhibitors during the study period. Strong inhibitors include: cobicistat; ritonavir; indinavir and ritonavir; itraconazole; ketoconazole; lopinavir and ritonavir; paritaprevir and ritonavir and ombitasvir (and/or dasabuvir); posaconazole; saquinavir and ritonavir; tipranavir and ritonavir; elvitegravir and ritonavir; telithromycin; voriconazole; ceritinib; clarithromycin; idealalisib; nefazodone; nelfinavir.
6. Subjects who are taking strong CYP3A4 Inducers within 14 days before the index procedure or plan to take the strong inducers during the study period. Strong inducers include apalutamide; carbamazepine; enzalutamide; ivosidenib; lumacaftor and ivacaftor; mitotane; phenytoin; rifampin; St. John's wort.

   * Angiographic Exclusion Criteria

Subject whose target lesion(s) meet any of the following angiographic criteria will be excluded from the trial:

1. Target lesion is totally occluded or has evidence of thrombus.
2. Target lesion is located in the left main or any arterial or venous graft.
3. Target lesion is in a side branch that is "jailed" by a main vessel stent.
4. In stent restenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure (TLF) | 12 months
  Target lesion failure (TLF) is defined as the composite of cardiac death, target-vessel myocardial infarction (MI) or clinically-driven target lesion revascularization (TLR) at 12 months.
  MI includes spontaneous (Type 1) MI using the 4th Universal Definition of Myocardial Infarction (UDMI) and peri-procedural MI using the Society for Cardiac Angiography and Intervention (SCAI) definition.
PK Sub-study Primary Endpoint 1 | 6 months
  PK parameters of C(max)
PK Sub-study Primary Endpoint 2 | 6 months
  PK parameters of T(max)
PK Sub-study Primary Endpoint 3 | 6 months
  PK parameters of AUC(last)
PK Sub-study Primary Endpoint 4 | 6 months
  PK parameters of MRT(last)

SECONDARY OUTCOMES:
Secondary Endpoint 1 | 12 months
  Composite of all-cause mortality, target vessel MI or clinically driven target lesion revascularization
Secondary Endpoint 2 | Up to 7 days
  Lesion success, defined as attainment of < 30% residual stenosis of target lesion using any percutaneous method
Secondary Endpoint 3 | Up to 7 days
  Procedure success, defined as attainment of < 30% residual stenosis of the target lesion using the assigned study device only without the occurrence of in-hospital major adverse cardiac events (MACE), composite of all-cause death, MI or any clinically-driven TLR.
Secondary Endpoint 4 | Up to 7 days and at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  Composite safety endpoint, defined as the patient-oriented composite of any death, any MI (spontaneous or peri-procedural), or any repeat revascularization.
Secondary Endpoint 5 | Up to 7 days and at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  All-Cause Mortality
Secondary Endpoint 6 | Up to 7 days and at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  Cardiovascular Mortality
Secondary Endpoint 7 | Up to 7 days and at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  MI (spontaneous MI using the 4th UDMI, peri-procedural MI using SCAI and Academic Research Consortium [ARC]-2 definitions)
Secondary Endpoint 8 | Up to 7 days and at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  Clinically-driven TLR
Secondary Endpoint 9 | Up to 7 days and at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  all TLR
Secondary Endpoint 10 | Up to 7 days and at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  Clinically-driven Target Vessel Revascularization (TVR)
Secondary Endpoint 11 | Up to 7 days and at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  all TVR
Secondary Endpoint 12 | Up to 7 days and at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  Non-target lesion revascularization
Secondary Endpoint 13 | Up to 7 days and at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  TLF
Secondary Endpoint 14 | Up to 7 days and at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  Target vessel failure (TVF), defined as a composite of: cardiac death, target vessel MI (spontaneous or peri-procedural) and any clinically-driven TVR
Secondary Endpoint 15 | Up to 7 days and at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  Stent or target lesion segment thrombosis (definite or probable) according to the ARC criteria for acute, subacute, late, very late and cumulative stent thrombosis
Secondary Endpoint 16 | 12 months
  Bleeding Academic Research Consortium (BARC) class 2-5
Secondary Endpoint 17 | Up to 7 days and at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  Net adverse clinical events, defined as death, MI (spontaneous or peri-procedural), TVR, stent/target lesion segment thrombosis or bleeding (BARC types 2-5, assessed to 12 months)

OTHER OUTCOMES:
PK Sub-Study Secondary Endpoint 1 | 6 months
  If calculations are valid, additional PK parameter of AUC(inf).
PK Sub-Study Secondary Endpoint 2 | 6 months
  If calculations are valid, additional PK parameter of Cl.
PK Sub-Study Secondary Endpoint 3 | 6 months
  If calculations are valid, additional PK parameter of Vz.
PK Sub-Study Secondary Endpoint 4 | 6 months
  If calculations are valid, additional PK parameter of Vss.
PK Sub-Study Secondary Endpoint 5 | 6 months
  If calculations are valid, additional PK parameter of half-life.
PK Sub-Study Secondary Endpoint 6 | 6 months
  Dose normalized C(max) will be considered if appropriate.
PK Sub-Study Secondary Endpoint 7 | 6 months
  Dose normalized AUC will be considered if appropriate.
PK Sub-Study Secondary Endpoint 8 | 6 months
  Device success, defined as attainment of ≤ 30% residual stenosis of the target lesion using the assigned device only

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute
Locations (43):
- United States (43):
  - St. Bernards, Jonesboro, Arkansas
  - CISD Sharp Chula Vista, Chula Vista, California
  - Cedars Sinai, Los Angeles, California
  - HCA Los Robles, Thousand Oaks, California
  - Harbor UCLA, Torrance, California
  - Colorado Heart and Vascular, Golden, Colorado
  - ClinRe, Thornton, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - HCA Florida JFK, Atlantis, Florida
  - Mease Countryside Hospital, Clearwater, Florida
  - University of Florida, Jacksonville, Jacksonville, Florida
  - HCA Largo, Largo, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Atlanta VA, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory, Atlanta, Georgia
  - Archbold Memorial Hospital, Thomasville, Georgia
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess, Boston, Massachusetts
  - Mass General, Boston, Massachusetts
  - Brigham & Women's, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Englewood Health, Englewood, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - NC Heart and Vascular, Raleigh, North Carolina
  - The Lindner Research Center at Christ, Cincinnati, Ohio
  - Penn State Health Hershey & Berks, Hershey, Pennsylvania
  - UPMC Pinnacle, Mechanicsburg, Pennsylvania
  - Lifespan Rhode Island & Miriam, Providence, Rhode Island
  - HCA Centennial, Nashville, Tennessee
  - Hendrick Health, Abilene, Texas
  - Baylor Scott and White - Dallas, Dallas, Texas
  - Medical City of Fort Worth, Fort Worth, Texas
  - Baylor Scott and White Plano, Plano, Texas
  - Baylor Scott and White - Temple, Temple, Texas
  - HCA Chippenham, Richmond, Virginia
  - Advocate Aurora St. Luke's, Milwaukee, Wisconsin